CLINICAL TRIAL: NCT00502437
Title: The Antigagging Effect of Granisetron (Kytril), an Antiemetic Drug, in Dental Situations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Model: Crossover | Masking: Double
Other Study IDs: 376-11.05.07HMO-CTIL
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2007-06

CONDITIONS: Antiggaging Effect; Antiemetic; Granisetron; Gag Reflex; Dental Situations
MeSH Terms: conditions — Gagging | interventions — Granisetron

INTERVENTIONS:
Drug: GRANISETRON

SUMMARY:
Antigagging effect of kytril (granisetron) an antiemetic drug in dental situations

Gagging in dental situations can be a problem to the patient and the operating dentist. There are not proven methods of eliminating this reflex which sometimes will not allow routine quality dental care.

Pharmacological and behavioral approaches to eliminate this reflex have been tried with limited success.

This suggested study will test a potent antiemetic drug used in other clinical situations such as antineoplastic treatment. Granisetron is a potential antagonist for the 5-hydroxytryptamine3-receptor - 5HT(3), The drug binds to the receptor and blocks the effect of nausea and vomiting. Kytril mechanism of action was successfully proven for various medical situations as a potential antiemetic agent. Our Center for dental sedation and anesthesia in the oral medicine department have received approval to use Granisetron as an antigagging drug in dental situations based on several pilot studies conducted in other medical centers in different clinical situations such as strabismus corrections, post hysterectomy and others. Our preliminary clinical impression is that pre-emptive IV administration of this drug to patients with increased gag reflex is beneficial.

In our research we try to investigate the possibility of using kytril in dental situations.

In the first stage of this research we will study the INTRAVENOUS use of this drug and its effects On normal subjects compare them to themselves with placebo. According to the results of this study we will go on to the second stage of the research and try the same drug under oral administration.

The purpose of this study is to test the antigagging effect of this drug in a controlled manner in dental situations.

Our working hypothesis is that administration of this drug in dental situations with success, will allow many patients to receive good dental care

ELIGIBILITY:
Inclusion Criteria:

* normal subjects

Exclusion Criteria:

* presence of systemic disease
* subjects under medication or drug or food complementary agents

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Eliezer Kaufman, DMD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel